CLINICAL TRIAL: NCT02917655
Title: PARQVE - Project Arthritis Recovering Quality of Life by Means of Education - A Prospective Randomized Study Comparing the Educational Program With and Without Multidisciplinary Care
Brief Title: P.A.R.Q.V.E III - Comparison of the Educational Program With and Without Multidisciplinary Care
Acronym: PARQVE3
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Marcia Uchoa Rezende, MD; PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 14833/16
Record Dates: First submitted 2016-07-07; First posted 2016-09-28 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2019-08

CONDITIONS: Osteoarthritis; Metabolic Diseases
Keywords: Education; Quality of Life; Osteoarthritis; Metabolic Syndrome
MeSH Terms: conditions — Osteoarthritis; Metabolic Diseases; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Educational Program Associated (EPA) (Experimental): 45 patients will participate in two days of lectures two-months apart on the subject of knee OA, but will also come to the hospital on months 1, 3 and 5 after the first class to consult about nutritional habits to be improved; on month 4 for a group therapy session with the psychologists, 7 sessions with the physical therapy team followed by 7 sessions with the physical educators team (once a week/4 weeks and once every two weeks, three times).
  Answer WOMAC, Lequesne, Numerical Rating Scales (NRS), IPAQ, Tampa Scale for Kinesiophobia (TSK); perform the STS30, TUG, six-minute test have calculated BMI and body fat percentage at baseline evaluations, 6, 12 and 24 months.
  Interventions: Behavioral: Womac; Behavioral: Lequesne; Behavioral: Numerical Rating Scales (NRS); Behavioral: IPAQ; Behavioral: STS30; Behavioral: TUG; Behavioral: Six-minute Test; Behavioral: Two days of lectures; Behavioral: Session with the psychologists; Behavioral: Sessions with the physical therapy team; Behavioral: Sessions with the physical educators team; Behavioral: Nutritional habits to be improved; Behavioral: Tampa Scale for Kinesiophobia (TSK)
- Educational Program Isolated (EPI) (Other): 45 patients will participate in two days of lectures two-months apart on the subject of knee OA.
  Answer WOMAC, Lequesne, Numerical Rating Scales (NRS), IPAQ, Tampa Scale for Kinesiophobia (TSK); perform the STS30, TUG, six-minute test have calculated BMI and body fat percentage at baseline evaluations, 6, 12 and 24 months.
  Interventions: Behavioral: Womac; Behavioral: Lequesne; Behavioral: Numerical Rating Scales (NRS); Behavioral: IPAQ; Behavioral: STS30; Behavioral: TUG; Behavioral: Six-minute Test; Behavioral: Two days of lectures; Behavioral: Tampa Scale for Kinesiophobia (TSK)

INTERVENTIONS:
Behavioral: Womac — Answer WOMAC at baseline, 6, 12 and 24 months.
Behavioral: Lequesne — Answer Lequesne at baseline, 6, 12 and 24 months.
Behavioral: Numerical Rating Scales (NRS) — Answer NRS at baseline, 6, 12 and 24 months.
Behavioral: IPAQ — Answer IPAQ at baseline, 6, 12 and 24 months.
Behavioral: STS30 — Perform the STS30 at baseline, 6, 12 and 24 months.
Behavioral: TUG — Perform the TUG at baseline, 6, 12 and 24 months.
Behavioral: Six-minute Test — Perform the six-minute test at baseline, 6, 12 and 24 months.
Behavioral: Two days of lectures — Participate in two days of classes about KOA, with the seven teams (orthopedics, psychology, physical therapy and fitness, occupational therapy, social workers and nutritionist).
Behavioral: Session with the psychologists — Participate in a extra session group with the psychology team about their experiences with the program
  Arms: Educational Program Associated (EPA)
Behavioral: Sessions with the physical therapy team — Participate in a extra session group with the physical therapists
  Arms: Educational Program Associated (EPA)
Behavioral: Sessions with the physical educators team — Participate in a extra session group with the physical educators
  Arms: Educational Program Associated (EPA)
Behavioral: Nutritional habits to be improved — Attend 3 extra meetings about nutrition.
  Arms: Educational Program Associated (EPA)
Behavioral: Tampa Scale for Kinesiophobia (TSK) — Answer Tampa Scale for Kinesiophobia (TSK) at baseline, 6 months, 12 and 24 months.

SUMMARY:
BACKGROUND: Osteoarthritis (OA), and particularly knee osteoarthritis (KOA) is a disorder that greatly impairs the quality of life of patients and its incidence increases with longevity, obesity and lower socioeconomic and educational level. It is expected that 40% of people over 60 have symptomatic OA of the knees and hips. The core treatment of OA is education, weight loss and increased physical activity. We create an educational program that improved function of the patients given by the sit-to-stand 30 seconds test (STS30). However, weight loss, an important foundation of clinical treatment, was only effective (more than 2 points in BMI) in 10% of the program participants. For greater effectiveness in weight loss and adherence to physical activity, we prepared an intensive program with more intensive nutritional care, psychological, physical therapy and physical trainers and compare the existing program educators. OBJECTIVE: To compare an educational program isolated to an educational program associated with nutritional consultations, group therapy sessions and progressed physiotherapy sessions to sessions with physical educators in patients with KOA and comorbidities (metabolic syndrome).

METHODS: Ninety patients with OAJ and co-morbidities (Two or more of: overweight or obesity, hyperglycemia, dyslipidemia, hyperuricemia, high blood pressure) will be divided into two groups: study (S) and control (C). Both groups will attend the two-day multi-professional classes on OA with two months interval. But the study group will also make three group consultations about nutrition, 1 extra session of group therapy with psychology team and 7 exercise sessions in groups with physical therapy and subsequently 7 sessions with physical educators. The groups will be evaluated for weight, height (to calculate BMI), waist-hip ratio, percentage of body fat, consumption of daily medications, WOMAC, Lequesne, IPAQ, Tampa Scale for Kinesiophobia (TSK), Sit to stand 30 seconds test (STS30), timed-up- and-go (TUG) and six minute test. At inclusion, six, twelve and 24 months after the classes.

DETAILED DESCRIPTION:
Given the inclusion criteria, patients undergo pre-evaluation by the multidisciplinary group composed of teams of orthopedic doctors, nutritionists, physical therapists, physical educators:

Orthopedics - it is treating the patients according to the guidelines of OARSI, offering everything we have for the treatment of OA at the Hospital das Clinicas.

Nutrition - It will measure the skinfold of all patients at baseline and at six and twelve months. As the draw, will attend the study group at 1, 3 and 5 months after the first class and the control group lose weight significantly less than the study group will meet the control group after one year in the same manner than has undergone the study group .

Physiotherapy - Undertake the test and sit ups, Timed-Up-and-Go (TUG) test and Sit to stand 30 seconds test (STS30) including six, twelve and 24 months after inclusion. The physiotherapy group will care study group sessions in a group of patients once a week for 4 weeks, 2 times a week for 1 month and 1x / month in the third month, giving exercises to be performed daily and charging them through the registration of patients. If the results of six and twelve months show better in the study group, the control group will do the same interventions the study group one year later.

Physical Education - will apply the questionnaire International Physical Activity Questionnaire, IPAQ, Tampa Scale for Kinesiophobia (TSK) and will make up test and down stairs and evaluating short version flexibility, inclusion, six, 12 and 24 months. After three months of exercise guided by physiotherapists, the study group will begin an exercise program with physical education teachers to become able to carry out alone or join a gym at the end of the sixth month of the program. It will also provide weekly classes for 1 month, biweekly in the second month and last month in the third charging the daily activities in the record of the patient's notebook.

ELIGIBILITY:
Inclusion Criteria:

* Men and women diagnosed with KOA with comorbidities (metabolic syndrome, ie, Osteoarthritis Knee + at least two of: overweight / obesity, hyperglycemia, dyslipidemia, hyperurecemia, hypertension, polyarthrosis) and up to 75 years old, capable of reading, understand and responding to the WOMAC questionnaire.
* Classified as stages I to III Kelgreen and Lawrence (K-L), i.e. without any degree of gonarthritis obliteration of joint space narrowing.
* With clinical treatment indication of OA.

Exclusion Criteria:

* Patients who have cognitive, and psychiatric or neurological disorders, whose symptoms during the evaluation are related to or significantly interfere in the functions of attention, memory, logical reasoning, understanding, interaction with the group, that would prevent assimilation of the given guidelines.
* Missing interventions

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
Evaluate function with the TUG (Time-up-Go test) | Baseline, 6, 12 and 24 months
  Apply TUG (Time-up-Go test) The data will be evaluated with absolute measures and changes in respect to baseline values at 6, 12 and 24 months.

SECONDARY OUTCOMES:
Evaluate improvement in pain | Baseline, 6, 12 and 24 months
  Apply the WOMAC questionnaire WOMAC (The Western Ontario and McMaster Universities Osteoarthritis Index)
Evaluate improvement in function | Baseline, 6, 12 and 24 months
  Apply the Lequesne questionnaire
Evaluate percentage of body fat. | Baseline, 6, 12 and 24 months
  Nine skinfolds measurements
Level of physical activity | Baseline, 6, 12 and 24 months
  Apply International Questionnaire physical activity Questionnaire-IPAQ short version.
Evaluate function with the STS30 (Sit to Stand 30 SecondsTest) | Baseline, 6, 12 and 24 months
  Apply STS30 (Sit to Stand 30 SecondsTest)
Evaluate the consumption of drugs | baseline to 6 months
  Both groups, starting from inclusion will record the daily consumption of drugs (baseline to 6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Marcia U Rezende, MD; PhD, Principal Investigator — Department of Orthopedics and Traumatology - Hospital das Clinicas da FMUSP

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lane NE, Brandt K, Hawker G, Peeva E, Schreyer E, Tsuji W, Hochberg MC. OARSI-FDA initiative: defining the disease state of osteoarthritis. Osteoarthritis Cartilage. 2011 May;19(5):478-82. doi: 10.1016/j.joca.2010.09.013. Epub 2011 Mar 23. PMID 21396464
- [Background] Woolf AD, Pfleger B. Burden of major musculoskeletal conditions. Bull World Health Organ. 2003;81(9):646-56. Epub 2003 Nov 14. PMID 14710506
- [Background] WHO Scientific Group on the Burden of Musculoskeletal Conditions at the Start of the New Millennium. The burden of musculoskeletal conditions at the start of the new millennium. World Health Organ Tech Rep Ser. 2003;919:i-x, 1-218, back cover. PMID 14679827
- [Background] Kwok WY, Vliet Vlieland TP, Rosendaal FR, Huizinga TW, Kloppenburg M. Limitations in daily activities are the major determinant of reduced health-related quality of life in patients with hand osteoarthritis. Ann Rheum Dis. 2011 Feb;70(2):334-6. doi: 10.1136/ard.2010.133603. Epub 2010 Nov 15. PMID 21081529
- [Background] Dawson J, Linsell L, Zondervan K, Rose P, Randall T, Carr A, Fitzpatrick R. Epidemiology of hip and knee pain and its impact on overall health status in older adults. Rheumatology (Oxford). 2004 Apr;43(4):497-504. doi: 10.1093/rheumatology/keh086. Epub 2004 Feb 3. PMID 14762225
- [Background] Dixon T, Shaw M, Ebrahim S, Dieppe P. Trends in hip and knee joint replacement: socioeconomic inequalities and projections of need. Ann Rheum Dis. 2004 Jul;63(7):825-30. doi: 10.1136/ard.2003.012724. PMID 15194578
- [Background] Mahomed NN, Barrett J, Katz JN, Baron JA, Wright J, Losina E. Epidemiology of total knee replacement in the United States Medicare population. J Bone Joint Surg Am. 2005 Jun;87(6):1222-8. doi: 10.2106/JBJS.D.02546. PMID 15930530
- [Background] Blagojevic M, Jinks C, Jeffery A, Jordan KP. Risk factors for onset of osteoarthritis of the knee in older adults: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2010 Jan;18(1):24-33. doi: 10.1016/j.joca.2009.08.010. Epub 2009 Sep 2. PMID 19751691
- [Background] Jorgensen KT, Pedersen BV, Nielsen NM, Hansen AV, Jacobsen S, Frisch M. Socio-demographic factors, reproductive history and risk of osteoarthritis in a cohort of 4.6 million Danish women and men. Osteoarthritis Cartilage. 2011 Oct;19(10):1176-82. doi: 10.1016/j.joca.2011.07.009. Epub 2011 Jul 27. PMID 21835256
- [Background] Zhang W, Moskowitz RW, Nuki G, Abramson S, Altman RD, Arden N, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis, Part II: OARSI evidence-based, expert consensus guidelines. Osteoarthritis Cartilage. 2008 Feb;16(2):137-62. doi: 10.1016/j.joca.2007.12.013. PMID 18279766
- [Background] Zhang W, Nuki G, Moskowitz RW, Abramson S, Altman RD, Arden NK, Bierma-Zeinstra S, Brandt KD, Croft P, Doherty M, Dougados M, Hochberg M, Hunter DJ, Kwoh K, Lohmander LS, Tugwell P. OARSI recommendations for the management of hip and knee osteoarthritis: part III: Changes in evidence following systematic cumulative update of research published through January 2009. Osteoarthritis Cartilage. 2010 Apr;18(4):476-99. doi: 10.1016/j.joca.2010.01.013. Epub 2010 Feb 11. PMID 20170770
- [Background] Bruyere O, Cooper C, Pelletier JP, Branco J, Luisa Brandi M, Guillemin F, Hochberg MC, Kanis JA, Kvien TK, Martel-Pelletier J, Rizzoli R, Silverman S, Reginster JY. An algorithm recommendation for the management of knee osteoarthritis in Europe and internationally: a report from a task force of the European Society for Clinical and Economic Aspects of Osteoporosis and Osteoarthritis (ESCEO). Semin Arthritis Rheum. 2014 Dec;44(3):253-63. doi: 10.1016/j.semarthrit.2014.05.014. Epub 2014 May 14. PMID 24953861
- [Background] McAlindon TE, Bannuru RR, Sullivan MC, Arden NK, Berenbaum F, Bierma-Zeinstra SM, Hawker GA, Henrotin Y, Hunter DJ, Kawaguchi H, Kwoh K, Lohmander S, Rannou F, Roos EM, Underwood M. OARSI guidelines for the non-surgical management of knee osteoarthritis. Osteoarthritis Cartilage. 2014 Mar;22(3):363-88. doi: 10.1016/j.joca.2014.01.003. Epub 2014 Jan 24. PMID 24462672
- [Background] Rosales Ade L, Brito NL, Frucchi R, de Campos GC, Pailo AF, de Rezende MU. Obesity, ostearthritis and clinical treatment. Acta Ortop Bras. 2014;22(3):136-9. doi: 10.1590/1413-78522014220300679. PMID 25061419
- [Background] Campos GC, Kohara MT, Rezende MU, Santana OF, Moreira MM, Camargo OP. Schooling of the patients and clinical application of questionnaires in osteoarthitis. Acta Ortop Bras. 2014;22(5):256-9. doi: 10.1590/1413-78522014220500980. PMID 25328433
- [Background] Shin D. Association between metabolic syndrome, radiographic knee osteoarthritis, and intensity of knee pain: results of a national survey. J Clin Endocrinol Metab. 2014 Sep;99(9):3177-83. doi: 10.1210/jc.2014-1043. Epub 2014 Apr 29. PMID 24780047
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Konstantinidis GA, Aletras VH, Kanakari KA, Natsis K, Bellamy N, Niakas D. Comparative validation of the WOMAC osteoarthritis and Lequesne algofunctional indices in Greek patients with hip or knee osteoarthritis. Qual Life Res. 2014 Mar;23(2):539-48. doi: 10.1007/s11136-013-0490-x. Epub 2013 Aug 6. PMID 23918463
- [Background] Shumway-Cook A, Brauer S, Woollacott M. Predicting the probability for falls in community-dwelling older adults using the Timed Up & Go Test. Phys Ther. 2000 Sep;80(9):896-903. PMID 10960937
- [Background] Britto RR, Probst VS, de Andrade AF, Samora GA, Hernandes NA, Marinho PE, Karsten M, Pitta F, Parreira VF. Reference equations for the six-minute walk distance based on a Brazilian multicenter study. Braz J Phys Ther. 2013 Nov-Dec;17(6):556-63. doi: 10.1590/S1413-35552012005000122. Epub 2013 Nov 14. PMID 24271092
- [Background] Sanghi D, Srivastava RN, Singh A, Kumari R, Mishra R, Mishra A. The association of anthropometric measures and osteoarthritis knee in non-obese subjects: a cross sectional study. Clinics (Sao Paulo). 2011;66(2):275-9. doi: 10.1590/s1807-59322011000200016. PMID 21484046
- See also: POF 2008-2009: desnutrição cai e peso das crianças brasileiras ultrapassa padrão internacional. — http://saladeimprensa.ibge.gov.br/noticias?busca=1&id=1&idnoticia=1699&t=pof-20082009-desnutricao-cai-peso-criancas-brasileiras-ultrapassa-padrao-internacional&view=noticia
- See also: PARQVE - Project Arthritis Recovering Quality of Life by means of Education. Short-term outcome in a randomized clinical trial — https://www.omicsonline.org/peer-reviewed/parqveproject-arthritis-recovering-quality-of-life-by-means-of-education-shortterm-outcome-in-a-randomized-clinical-trial-20432.html
- See also: Prevalence and incidence of hand osteoarthritis and upper limb complaints in patients with knee osteoarthritis .... in a educational osteoarthritis program — http://www.scirp.org/journal/PaperInformation.aspx?paperID=62765
- See also: Analysis of anthropometric measurements and dietary intake in patients undergoing a multi-professional ostearthritis education program (PARQVE - Project Arthritis Recovering Quality of Life by means of Education) — http://www.scirp.org/journal/PaperInformation.aspx?PaperID=63851